CLINICAL TRIAL: NCT03727945
Title: Posture Correction in Abdominopelvic Training in Women With Stress Urinary Incontinence
Brief Title: Posture in Abdominopelvic Training in Women SUI
Acronym: QoL SUI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Laura Fuentes Aparicio, PhD Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H1410616852782,
Record Dates: First submitted 2018-10-28; First posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Female Stress Incontinence
Keywords: stress urinary incontinence; abdominopelvic exercise; quality of life
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Posture

STUDY DESIGN:
Intervention Model Description: 2 aleatorized groups; control group (n=21) and intervention group
Who Masked: Participant
Masking Description: Urolog was not involved in physiotherapy treatment, randomised patients previous of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- abdominopelvic exercise and posture (Experimental): N=21 received supervised physiotherapy abdominopelvic exercise previous postural correction.
  Interventions: Other: abdominopelvic exercise and posture
- abdominopelvic exercise (Experimental): N=21 received supervised physiotherapy abdominopelvic exercise.
  Interventions: Other: abdominopelvic exercise

INTERVENTIONS:
Other: abdominopelvic exercise and posture — n=21 women received supervised abdominopelvic exercise with previous postural correction. During 12 sessions a specialized physiotherapist supervised to realization of progressive abdominopelvic exercises, previous explain postural correction pelvis, cervical and dorsal zone.
  Arms: abdominopelvic exercise and posture
Other: abdominopelvic exercise — n=21 women received supervised abdominopelvic exercise. During 12 sessions a specialized physiotherapist supervised to realization of progressive abdominopelvic exercises.
  Arms: abdominopelvic exercise

SUMMARY:
Measure effect of postural correction in abdominopelvic exercises on the improvement of the quality of life in patients with SUI. 42 women aged between 46-75 with SUI and stress-predominant mixed urinary incontinence. There were randomly assigned two groups of different treatment.

Quality of life was measured by questionnaires: Incontinence Questionnaire Short Form (ICIQ-IU-SF) and King's Health Questionnaire (KHQ) global punctuation and incontinence impact. Treatment satisfaction was measured by VAS scale.

DETAILED DESCRIPTION:
The aim of this study was compare the effect of postural correction in abdominopelvic exercises on the improvement of the quality of life in patients with stress urinary incontinence (SUI).

Was a randomized 2-treatment parallel design study. The sample consist in 42 women aged between 46-75 with stress urinary incontinence (SUI) and stress-predominant mixed urinary incontinence (IUM). They were randomly assigned to two groups: Group 1 (n=21) who received abdomino-pelvic training, and Group 2(n=21) who received the above treatment, guidelines about postural correction.

Both groups received 12 treatment sessions in first session information regarding clinical and demographical aspects will be collected.

To evaluate results of postural correction combined with abdominopelvic exercise women was assessed:at initial session, post- intervention and 3 months post-intervention treatment.Quality of life was measured by spanish validation questionnaires: International Continence Questionnaire Short Form (ICIQ-IU-SF) and King's Health Questionnaire (KHQ) global punctuation and incontinence impact. Treatment satisfaction was measured by Visual analogic scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* SUI or stress-predominant mixed UI
* diagnosed via clinical assessment and urodynamic study
* Estrogenic deficit.: perimenopause, menopause, postmenopause

Exclusion Criteria:

* grade 3-4 prolapse,
* functional alterations (Barthel Scale > 85 points),
* neurological or cognitive alterations (mini mental examination > 24 points)
* other predominant type of urinary incontinence.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 45-75 years and hormonal state
Enrollment: 49 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Changes from Quality of life. KHQ | baseline,3 months,6 months
  The questionnaire KHQ consists of 30 items distributed in 9 dimensions that we expose below, the scores of this questionnaire vary from 0 to 100, each item presents a scale type Likert with four options of response. The score of the KHQ questionnaire can be globally with a range of 0 (which indicates better health-related quality of life) at 100 points (indicating a worse quality of life)
Changes from Quality of life. ICIQ-IU-SF | baseline,3 months, 6 months
  t consists of four questions that assess the presence of urge urinary incontinence, the amount of fluid evacuated and the involvement of the quality of life. The final score oscillates from 0-21, indicating higher scores to greater severity of the IU.
Treatment satisfaction | 3 months
  Visual analogic scale (VAS, 0-10, 0=minimum score, 10=maximum score). Higher values represent a better outcome (less treatment satisfaction)
Changes from IU impact. KHQ | baseline,3 months, 6 months
  Question nº2 of KHQ measured IU impact in patient's life. Is a Likert scale 0-4 punctuation ( 0= no proceed, 4= A lot)
Changes from IU impact.ICIQ-IU-SF | Initial,3 months, 6 months
  Question nº3 of ICIQ-IU-SF, measured IU impact in patient's life.Is a numeric scale (1-10),(1= none and 10= a lot )

IPD SHARING:
Plan to Share IPD: Undecided
The fist idea was make a Doctoral Thesis. But the investigators continue investigating in this area.

REFERENCES:
- [Background] 1. Salinas Casado J, Díaz Rodríguez A, Brenes Bermúdez F, Cancelo Hidalgo MJ, Cuenllas Díaz A, Verdejo Bravo C. Prevalencia de la incontinencia urinaria en España. UROD A. 2010; 23 (1): 52-66. 2. Aguilar-Navarro SG, Incontinencia urinaria en el adulto mayor. Rev Enferm Inst Mex Seguro Soc. 2007; 15 (1): 51-56. 3. Zunzunegui Pastor MV, Rodríguez Laso A, García de Yébenes MJ, Aguilar Conesa M.D, Lázaro y de Mercado P y Otero Puime A. Prevalencia de la incontinencia urinaria y factores asociados en varones y mujeres de más de 65 años. Aten Primaria. 2003; 32 (6): 337-342. 4. Grosse D, Sengler J. Reeducación del periné fisioterapia en las incontinencias urinarias. Ed Masson. 2001. 5. Robles JE (editor). I Curso de formación en incontinencia urinaria. Pamplona: Newbook ediciones. 2001. 6. Guía clínica sobre la incontinencia urinaria. Schroder A, Abrams P. Andersson KE, Artibani W, Chapple CR, Drake MJ, Hampel C, Neisius A, Tubaro A, Thuroff JW. European Association of Urology. 2010. 7. Lacima G, Espuña M. Patología del suelo pélvico. Gastroenterol Hepatol. 2008; 31 (9): 587-595. 8. Sapsford R. The pelvic floor. A clinical model for function and rehabilitation. Physiotherapy. 2001; 87 (12): 620-630.